CLINICAL TRIAL: NCT03009318
Title: Combination of 11C-MET PET and MRS in the Diagnosis of Glioma.
Brief Title: MRS and 11C-methionine PET/CT in the Diagnosis of Glioma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Dongxiao Zhuang, Professor, Huashan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 81171295
Record Dates: First submitted 2016-12-29; First posted 2017-01-04 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Glioma
Keywords: Glioma; Magnetic resonance spectroscopy; Methionine; PET/CT
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MRS imaging and 11C-MET PET/CT (Other): Each patient underwent both MRS and MET PET before surgery.
  Interventions: Other: tumors are confirmed by surgery and pathology

INTERVENTIONS:
Other: tumors are confirmed by surgery and pathology — Each patient undergoes both MRS and MET PET scan before surgery. The lesion will be considered as a glioma when either MRS or MET PET results indicated the diagnosis. Pathologic diagnosis will be performed to confirm the final diagnosis.

SUMMARY:
MET PET and MRS are often performed as imaging tool for the differential diagnosis of gliomas. But both techniques have limitations causing misdiagnosis; thus, the investigators tried to combine these two imaging tools to study whether the combination of MET PET and MRS could raise the diagnosis ability of the radiological diagnosis of gliomas.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with non-enhancing supratentorial lesions shown by contrast-enhanced MRI
2. No surgery, chemotherapy or radiotherapy history
3. All patients gave written informed consent.

Exclusion Criteria:

1. Patients with infratentorial Neoplasms
2. Patients with enhancing supratentorial lesions
3. Recurrent gliomas after surgery
4. Primary gliomas with history of radiotherapy or chemotherapy
5. History of malignant tumours at any body site
6. Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-01; Primary Completion 2016-09 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Sensitivity of the combination of MRS and 11C-MET PET/CT | 5 years

SECONDARY OUTCOMES:
The relationship between 11C-MET PET/CT results and molecular pathogeneses | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Dongxiao Zhuang, Professor, Principal Investigator — Huashan Hospital, Sudan University
Locations (1):
- Huashan hospital, Fudan university, Shanghai, China

REFERENCES:
- [Background] Ostrom QT, Gittleman H, Liao P, Rouse C, Chen Y, Dowling J, Wolinsky Y, Kruchko C, Barnholtz-Sloan J. CBTRUS statistical report: primary brain and central nervous system tumors diagnosed in the United States in 2007-2011. Neuro Oncol. 2014 Oct;16 Suppl 4(Suppl 4):iv1-63. doi: 10.1093/neuonc/nou223. No abstract available. PMID 25304271
- [Background] Fouke SJ, Benzinger T, Gibson D, Ryken TC, Kalkanis SN, Olson JJ. The role of imaging in the management of adults with diffuse low grade glioma: A systematic review and evidence-based clinical practice guideline. J Neurooncol. 2015 Dec;125(3):457-79. doi: 10.1007/s11060-015-1908-9. Epub 2015 Nov 3. PMID 26530262
- [Background] Wang W, Hu Y, Lu P, Li Y, Chen Y, Tian M, Yu L. Evaluation of the diagnostic performance of magnetic resonance spectroscopy in brain tumors: a systematic review and meta-analysis. PLoS One. 2014 Nov 13;9(11):e112577. doi: 10.1371/journal.pone.0112577. eCollection 2014. PMID 25393009
- [Background] Martinez-Bisbal MC, Celda B. Proton magnetic resonance spectroscopy imaging in the study of human brain cancer. Q J Nucl Med Mol Imaging. 2009 Dec;53(6):618-30. PMID 20016453
- [Background] Guo J, Yao C, Chen H, Zhuang D, Tang W, Ren G, Wang Y, Wu J, Huang F, Zhou L. The relationship between Cho/NAA and glioma metabolism: implementation for margin delineation of cerebral gliomas. Acta Neurochir (Wien). 2012 Aug;154(8):1361-70; discussion 1370. doi: 10.1007/s00701-012-1418-x. Epub 2012 Jun 23. PMID 22729482
- [Background] Yamasaki F, Takayasu T, Nosaka R, Amatya VJ, Doskaliyev A, Akiyama Y, Tominaga A, Takeshima Y, Sugiyama K, Kurisu K. Magnetic resonance spectroscopy detection of high lipid levels in intraaxial tumors without central necrosis: a characteristic of malignant lymphoma. J Neurosurg. 2015 Jun;122(6):1370-9. doi: 10.3171/2014.9.JNS14106. Epub 2015 Mar 6. PMID 25748300
- [Background] Oz G, Alger JR, Barker PB, Bartha R, Bizzi A, Boesch C, Bolan PJ, Brindle KM, Cudalbu C, Dincer A, Dydak U, Emir UE, Frahm J, Gonzalez RG, Gruber S, Gruetter R, Gupta RK, Heerschap A, Henning A, Hetherington HP, Howe FA, Huppi PS, Hurd RE, Kantarci K, Klomp DW, Kreis R, Kruiskamp MJ, Leach MO, Lin AP, Luijten PR, Marjanska M, Maudsley AA, Meyerhoff DJ, Mountford CE, Nelson SJ, Pamir MN, Pan JW, Peet AC, Poptani H, Posse S, Pouwels PJ, Ratai EM, Ross BD, Scheenen TW, Schuster C, Smith IC, Soher BJ, Tkac I, Vigneron DB, Kauppinen RA; MRS Consensus Group. Clinical proton MR spectroscopy in central nervous system disorders. Radiology. 2014 Mar;270(3):658-79. doi: 10.1148/radiol.13130531. PMID 24568703
- [Background] WRENN FR Jr, GOOD ML, HANDLER P. The use of positron-emitting radioisotopes for the localization of brain tumors. Science. 1951 May 4;113(2940):525-7. doi: 10.1126/science.113.2940.525. No abstract available. PMID 14828392
- [Background] Demetriades AK, Almeida AC, Bhangoo RS, Barrington SF. Applications of positron emission tomography in neuro-oncology: a clinical approach. Surgeon. 2014 Jun;12(3):148-57. doi: 10.1016/j.surge.2013.12.001. Epub 2014 Mar 11. PMID 24629841
- [Background] Herholz K, Holzer T, Bauer B, Schroder R, Voges J, Ernestus RI, Mendoza G, Weber-Luxenburger G, Lottgen J, Thiel A, Wienhard K, Heiss WD. 11C-methionine PET for differential diagnosis of low-grade gliomas. Neurology. 1998 May;50(5):1316-22. doi: 10.1212/wnl.50.5.1316. PMID 9595980
- [Background] Kracht LW, Miletic H, Busch S, Jacobs AH, Voges J, Hoevels M, Klein JC, Herholz K, Heiss WD. Delineation of brain tumor extent with [11C]L-methionine positron emission tomography: local comparison with stereotactic histopathology. Clin Cancer Res. 2004 Nov 1;10(21):7163-70. doi: 10.1158/1078-0432.CCR-04-0262. PMID 15534088
- [Background] Glaudemans AW, Enting RH, Heesters MA, Dierckx RA, van Rheenen RW, Walenkamp AM, Slart RH. Value of 11C-methionine PET in imaging brain tumours and metastases. Eur J Nucl Med Mol Imaging. 2013 Apr;40(4):615-35. doi: 10.1007/s00259-012-2295-5. Epub 2012 Dec 12. PMID 23232505